CLINICAL TRIAL: NCT01202344
Title: Computer Prediction of Restenosis Following Peripheral Angioplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: Dheeraj Rajan (Other)
Responsible Party: Sponsor-Investigator, Dheeraj Rajan, Associate Professor, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-0335-BE
Record Dates: First submitted 2010-09-10; First posted 2010-09-15 (Estimated); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Peripheral Angioplasty
Keywords: Angioplasty; Stenosis; Restenosis; Elastic Recoil; cheduled for percutaneous dilation of a peripheral artery; Target lesion in native artery; Baseline lumen diameter greater than 4 mm
MeSH Terms: conditions — Constriction, Pathologic

ARMS (2):
- Restenosis (Other): Patients who have restinosis immediately following angioplasty.
  Interventions: Other: Additional x-ray images
- No Restenosis (Other): Patients who do not have restinosis immediately following angioplasty.
  Interventions: Other: Additional x-ray images

INTERVENTIONS:
Other: Additional x-ray images — Approximately 3 additional x-ray images following angioplasty (within 1 hour)

SUMMARY:
The purpose of this study is to develop a computer program that might be able to accurately assess the risk of artery re-narrowing following angioplasty or stenting based on computer images. After angioplasty (a procedure to re-open narrowed or blocked blood vessels) the patients will have extra images taken in order to assess the results of the procedure; which will then be used to see whether or not these images can help predict outcomes such as the patient having to come back to the hospital to have the procedure done again.

DETAILED DESCRIPTION:
The study involves medical imaging of patients undergoing an angioplasty intervention in a peripheral artery. It is similar to an observational study, except that additional imaging is performed which is above the standard-of-care. Some risks may be associated with the additional imaging due to a small increase in radiation exposure and intravenous contrast administration. No investigational drug or device will be tested in this study. No control group will be used.

Logistic regression analysis will be performed using NCSS statistical software to identify which explanatory variable(s), selected from the simulation results, can be used to predict binary restenosis, the categorical dependent variable.

For each subject, binary restenosis will be determined by comparing the CT-scan images obtained 1 hour post-intervention to those obtained at the 6 month follow-up study. The CT-scan images will be segmented and a mesh of the target vessel will be reconstructed as described in objective 1. The lumen area will be measured in every cross-section of the mesh perpendicular to the vessel centerline, with 2 mm steps between cross-sections. The minimum lumen diameter will be calculated from the minimum lumen area. If the minimum lumen diameter at follow-up is less than 50% of the minimum lumen diameter post-intervention, then the binary restenosis is positive. Otherwise it is negative.

Objective 1: Evaluate the accuracy of computer predictions of artery dilatation and stent implantation from CT-scan images. This information is hypothesized to be indicative of the accuracy of other quantities predicted by computer simulation of angioplasty, such as those used as independent variables in objective 2.

Objective 2: Establish a regression model with 80% sensitivity and 80% specificity for predicting binary restenosis based on one or several injury parameters in patients undergoing angioplasty. The candidate injury parameters are:

* endothelium denudation (in % of total endothelium area)
* descriptors of the magnitude and spatial distribution of stretch ratio in the arterial wall
* descriptors of the magnitude and spatial distribution of intramural stress in the arterial wall All injury parameters are predicted by computer simulation of angioplasty.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for percutaneous dilation of a peripheral artery;
* age more than 18 years;
* informed consent signed by the subject;
* target lesion in native artery;
* baseline lumen diameter greater than 4 mm.

Exclusion Criteria:

* previous revascularization of the target lesion;
* subject undergoing chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-09; Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Simulation Accuracy | less than 6 hours after the procedure
  From the pre-intervention CT-scans, the target artery, calcium and lumen will be segmented, meshed and used to simulate the angioplasty steps. Simulation accuracy will be evaluated by comparing geometrical descriptors of the artery and lumen size and shape calculated in the simulation to those measured on the post-intervention CT scan images.

SECONDARY OUTCOMES:
Logistic Regression Analysis | 6 months
  Logistic regression analysis will be performed using NCSS statistical software to identify which explanatory variable(s), selected from the simulation results, can be used to predict binary restenosis, the categorical dependent variable.
  Binary restenosis will be determined by comparing the CT-scan images obtained 1 hour post-intervention to those obtained at the 6 month follow-up study.

CONTACTS AND LOCATIONS:
Overall Officials: Dheeraj Rajan, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Background] Hoffmann R, Mintz GS, Mehran R, Kent KM, Pichard AD, Satler LF, Leon MB. Tissue proliferation within and surrounding Palmaz-Schatz stents is dependent on the aggressiveness of stent implantation technique. Am J Cardiol. 1999 Apr 15;83(8):1170-4. doi: 10.1016/s0002-9149(99)00053-3. PMID 10215278
- [Background] Koyama J, Owa M, Sakurai S, Shimada H, Hikita H, Higashikata T, Ikeda S. Relation between vascular morphologic changes during stent implantation and the magnitude of in-stent neointimal hyperplasia. Am J Cardiol. 2000 Oct 1;86(7):753-8. doi: 10.1016/s0002-9149(00)01075-4. PMID 11018195
- [Background] Syeda B, Wexberg P, Gyongyosi M, Denk S, Beran G, Kiss K, Sperker W, Glogar D. Effects of radial stretch on target lesion revascularization after percutaneous coronary intervention: an intravascular ultrasound study. Can J Cardiol. 2003 May;19(6):691-7. PMID 12772020
- [Background] Schwartz RS, Huber KC, Murphy JG, Edwards WD, Camrud AR, Vlietstra RE, Holmes DR. Restenosis and the proportional neointimal response to coronary artery injury: results in a porcine model. J Am Coll Cardiol. 1992 Feb;19(2):267-74. doi: 10.1016/0735-1097(92)90476-4. PMID 1732351
- [Background] Rogers C, Tseng DY, Squire JC, Edelman ER. Balloon-artery interactions during stent placement: a finite element analysis approach to pressure, compliance, and stent design as contributors to vascular injury. Circ Res. 1999 Mar 5;84(4):378-83. doi: 10.1161/01.res.84.4.378. PMID 10066671
- [Background] Capron L, Bruneval P. Influence of applied stress on mitotic response of arteries to injury with a balloon catheter: quantitative study in rat thoracic aorta. Cardiovasc Res. 1989 Nov;23(11):941-8. doi: 10.1093/cvr/23.11.941. PMID 2611802
- [Background] Olson NE, Chao S, Lindner V, Reidy MA. Intimal smooth muscle cell proliferation after balloon catheter injury. The role of basic fibroblast growth factor. Am J Pathol. 1992 May;140(5):1017-23. PMID 1580326
- [Background] Jamal A, Bendeck M, Langille BL. Structural changes and recovery of function after arterial injury. Arterioscler Thromb. 1992 Mar;12(3):307-17. doi: 10.1161/01.atv.12.3.307. PMID 1547190
- [Background] Doornekamp FN, Borst C, Post MJ. Endothelial cell recoverage and intimal hyperplasia after endothelium removal with or without smooth muscle cell necrosis in the rabbit carotid artery. J Vasc Res. 1996 Mar-Apr;33(2):146-55. doi: 10.1159/000159143. PMID 8630348
- [Background] Nugent HM, Rogers C, Edelman ER. Endothelial implants inhibit intimal hyperplasia after porcine angioplasty. Circ Res. 1999 Mar 5;84(4):384-91. doi: 10.1161/01.res.84.4.384. PMID 10066672